CLINICAL TRIAL: NCT01712087
Title: Long-term Surveillance of the MedStream Programmable Infusion System for the Intrathecal Infusion of Baclofen in the Treatment of Spasticity
Brief Title: Long-term Surveillance of the MedStream Programmable Infusion System
Status: Terminated | Type: Observational
Why Stopped: Lack of enrollment
Sponsor: Codman & Shurtleff (Industry)
Responsible Party: Sponsor
Other Study IDs: NM-PMK-1001
Record Dates: First submitted 2012-10-19; First posted 2012-10-23 (Estimated); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Spasticity
Keywords: spasticity; muscle spasticity; muscle rigidity; motor neuron disease; hyperreflexia
MeSH Terms: conditions — Muscle Spasticity; Muscle Rigidity; Motor Neuron Disease; Reflex, Abnormal

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- MedStream System Implants: All subjects presenting for a de novo programmable pump implant or replacement of an implantable, programmable infusion pump for the treatment of severe spasticity with intrathecal Baclofen.
  Interventions: Device: MedStream Programmable Infusion System

INTERVENTIONS:
Device: MedStream Programmable Infusion System — Intrathecal Infusion of Baclofen in the Treatment of Spasticity
  Other Names: MedStream; MedStream Pump; MedStream programmable pump; MedStream Intrathecal Infusion System; MedStream Infusion system

SUMMARY:
This post-approval study will primarily evaluate the long-term safety of the MedStream Programmable Infusion System when used in combination with Baclofen for the treatment of severe spasticity. A secondary objective, to assess long-term effectiveness, based on the observed scores on the Ashworth Scale (rigidity for the lower extremities) and their Spasm Scores over the 36-month follow-up period will also be described.

ELIGIBILITY:
Inclusion Criteria:

* The subject is a viable candidate for "de novo" or continued (pump replacement) therapy for the treatment of severe spasticity with intrathecal Baclofen delivered by an implantable programmable pump.
* The subject or his/her Legally Authorized Representative must voluntarily provide Informed Consent for participation in this study in accordance with 21 Code of Federal Regulations (CFR) Part 50.
* The subject is willing to comply with the protocol-specified follow-up visit requirements for a period of 36 months after implant.
* The subject has an anticipated life expectancy of 24 months or greater.
* The subject must be 18 years of age or older at time of MedStream implant procedure.
* The subject is of sufficient body size to accommodate pump placement, in the opinion of the Investigator.
* The subject will receive a de novo or replacement implant of the MedStream 20 mL or 40 mL pump, MedStream approved catheter(s) and MedStream accessories.
* The Investigator intends to use Baclofen in the pump for treatment of severe spasticity
* The subject is capable of self-reporting spasm frequency.

Exclusion Criteria:

* Concurrent enrollment in an investigational device or drug study that has not completed the required follow-up period.
* Subject has had an infection and/or inflammation at or near the pump and/or catheter implantation site(s) within 30 days preceding enrollment.
* Evidence of a fever or infection within 10 days prior to the surgical implant procedure that, in the opinion of the Investigator might impact a successful pump implant.
* The subject has known hypersensitivity/allergies or contraindication to Baclofen or the materials in the infusion pump or catheter(s).
* The subject has a co-morbid condition that could limit his/her ability to participate in the study or to comply with the follow-up requirements or, which might impact the scientific integrity of the study.
* The subject has a rapid degenerative neurological disease such as lateral sclerosis, amyotrophic lateral sclerosis (ALS), rapidly progressive Multiple Sclerosis, inherited or rapidly progressive leukodystrophies, Moyamoya disease, cerebral autosomal dominant arteriopathy with subcortical infarcts and leucoencephalopathy (CADASIL), thrombophilias, rapidly progressive autoimmune disorders, or any disorder where progression of the underlying spinal cord or a central nervous system (CNS) disease is expected to progress significantly over the next 3 years
* Subject is a prisoner.
* Subject was previously enrolled in this study.
* Subject is pregnant or breastfeeding. (Note: females of child bearing potential must have a negative pregnancy test prior to enrollment in the study).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects presenting for a de novo programmable pump implant or replacement of an implantable, programmable infusion pump for the treatment of severe spasticity with intrathecal Baclofen are potential study candidates and will be screened for study eligibility. Subjects who do not meet all inclusion/exclusion criteria will not be enrolled into this study.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2012-10-01 (Actual); Primary Completion 2017-12-17 (Actual); Study Completion 2017-12-17 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the incidence of MedStream system-related Adverse Events (AE) | 24 Months
  The primary endpoint is the incidence of MedStream system-related AEs (MedStream pump and catheters) based on Clinical Events Committee determination of relationship, that occur from the start of the MedStream implant procedure (incision) until completion of the 24 month follow-up visit

SECONDARY OUTCOMES:
MedStream system-related AEs occurring from 24 to 36 months | 36 Months
Device-related AEs occurring with both MedStream and non-MedStream devices used or implanted during the course of the study. | 24 Months
  Device-related AEs occurring in subjects with both MedStream and non-MedStream devices used or implanted during the course of the study. Device refers to the pump and intrathecal catheters
Procedure-related AEs | 24 Months
  Procedure-related AEs including, but not limited to the following study procedures: MedStream system implant, pump refill and bolus, and reprogramming. If non-MedStream devices or components are utilized in these procedures, this will be described.
Drug-related AEs associated with intrathecal Baclofen | 24 Months
Drug-related AEs associated with other intrathecally-administered medications | 24 Months
Disease-related AEs associated with pre-existing conditions | 24 Months
  Disease-related AEs associated with pre-existing conditions that demonstrate a significant worsening of the disease or an increase in the frequency of episodes since baseline, as determined by the investigator.
Serious Adverse Events (SAEs) | 36 Months
Unanticipated Adverse Device Effects (UADEs) | 24 Months
The secondary effectiveness endpoints will be long-term effectiveness of MedStream System | 24 Month
  Long-term effectiveness as demonstrated by scores on the Ashworth Scale (lower extremity) and the frequency and severity components of the Penn Spasm Frequency Scale (PSFS) measured pre-implant, post-implant and at each of the protocol-specified study visits.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan T Megerian, MD, Study Director — Codman & Shurtleff
Locations (2):
- United States (2):
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - Methodist Hospital Research Institute, Houston, Texas